CLINICAL TRIAL: NCT00690469
Title: Carcinogen Metabolism, DNA Repair, Parental Exposures and Retinoblastoma
Brief Title: Genetic Mutations and Environmental Exposure in Young Patients With Retinoblastoma and in Their Parents and Young Healthy Unrelated Volunteers
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AEPI05N1; NCI-2009-00366 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-AEPI05N1; CDR0000588296; AEPI05N1; AEPI05N1 (Other: Childrens Oncology Group); AEPI05N1 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2008-06-03; First posted 2008-06-04 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2018-07

CONDITIONS: Extraocular Retinoblastoma; Intraocular Retinoblastoma; Recurrent Retinoblastoma
MeSH Terms: conditions — Retinoblastoma

GROUPS / COHORTS (1):
- Observational (biomarker analysis): Participants undergo a structured telephone interview questionnaire. The parental questionnaires collect basic demographic data (including age, race, education, and income), occupational history, medical radiation exposure, diet and supplement use (for the year before pregnancy for father, during pregnancy for mother), tobacco use, and alcohol use. The mothers are also asked about residential pesticides and prior assisted reproductive technology.
  Controls (parents) provide saliva samples. If a patient is also enrolled on COG-ARET0332, then the patient blood and tumor samples should be submitted. Parents of patients on this protocol should also submit a blood sample. Blood samples from the affected child, and blood and/or sputum samples from the parents may be submitted. Tumor specimens should be submitted if available.
  For some patients, a RB1 mutation detection assay on DNA derived from peripheral blood is performed. If the mutation is found, the parents? DNA is also screened.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This laboratory study is looking at genetic mutations and environmental exposure in young patients with retinoblastoma and in their parents and young healthy unrelated volunteers. Gathering information about gene mutations and environmental exposure may help doctors learn more about the causes of retinoblastoma in young patients.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To investigate the role of genotypes for carcinogen metabolizing enzymes (CME) and DNA repair proteins(DRPs) of the father of children diagnosed with retinoblastoma (RB) and his environmental exposures prior to the child?s conception in the etiology of sporadic bilateral retinoblastoma.

II. To test if the prevalence of preconception environmental exposures and polymorphisms with known or predicted functional consequences in genes for CMEs and DRPs is different in fathers of children with sporadic bilateral RB compared with fathers of the control group.

III. To test if the prevalence of the father?s preconception environmental exposures and his polymorphisms in CMEs and DRPs differs between subsets of cases defined by the type of mutation at the RB1 gene locus.

IV. To investigate the role of genotypes for CMEs and DRPs of the mother and child and environmental exposures after the child?s conception in the etiology of sporadic unilateral RB.

V. To test if the prevalence of environmental exposures during the pregnancy and polymorphisms with known or predicted functional consequences in CMEs is different in the mothers of children with sporadic unilateral RB compared with mothers of the control group.

VI. To test if the prevalence of polymorphisms in genes for CMEs and DRPs with known or predicted functional consequences is different in the children with sporadic unilateral RB compared with controls.

VII. To test if the prevalence of gestational exposures and polymorphisms in genes for CMEs of the mother and the polymorphisms in genes for CME and DRPs in the children differs between subsets of cases defined by the type of mutation at the RB1 gene locus.

OUTLINE: This is a multicenter study.

Participants undergo a structured telephone interview questionnaire. The parental questionnaires collect basic demographic data (including age, race, education, and income), occupational history, medical radiation exposure, diet and supplement use (for the year before pregnancy for father, during pregnancy for mother), tobacco use, and alcohol use. The mothers are also asked about residential pesticides and prior assisted reproductive technology.

Controls (parents) provide saliva samples. If a patient is also enrolled on COG-ARET0332, then the patient blood and tumor samples should be submitted. Parents of patients on this protocol should also submit a blood sample. Blood samples from the affected child, and blood and/or sputum samples from the parents may be submitted. Tumor specimens should be submitted if available.

For some patients, a RB1 mutation detection assay on DNA derived from peripheral blood is performed. If the mutation is found, the parents? DNA is also screened. Blood samples undergo DNA-based sequencing analysis, single nucleotide polymorphism genotyping, quantitative Southern blot analysis, isolation of RNA and reverse transcriptase-polymerase chain reaction analysis, and loss of heterozygosity analysis.

ELIGIBILITY:
Inclusion Criteria:

* Cases must meet the following criteria:

  * Diagnosed with sporadic retinoblastoma (RB) on or after 07/01/2006

    * No familial retinoblastoma
  * Have permission of physician to contact the parents
  * Diagnosed and/or treated at a Children's Oncology Group (COG) institution or *Wills Eye Hospital
* Controls must meet 1 of the following criteria:

  * Mother of a child with unilateral RB
  * Father of a child with bilateral RB
  * Age-matched non-blood-related child if possible
* Must reside in the U.S. or Canada
* Must have telephone in the home
* Biological parent speaks English or Spanish
* Concurrent treatment on a therapeutic trial is NOT required

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2008-06-02 (Actual); Primary Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
Association of the probability of having a child with bilateral retinoblastoma (RB) with the paternal genotype for selected DNA repair and carcinogen metabolizing enzymes (CME) genes | Not Provided
Probability that mothers of unilateral RB cases are more likely to have specific DNA-repair gene variants than the mothers of the control group | Not Provided
Significant effect of specific DNA repair and CME genotypes on the risk of unilateral RB | Not Provided
Probability that the bilateral RB1 mutation subtype will vary by DNA repair or CME genotype or preconception exposures of the fathers of bilateral RB cases | Not Provided
Probability that the unilateral RB1 mutation subtype will vary by DNA repair or CME genotype of the mother, of the affected child, and with gestational exposures | Not Provided

CONTACTS AND LOCATIONS:
Overall Officials: Greta Bunin, Principal Investigator — Children's Oncology Group
Locations (52):
- United States (49):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia Regional, Columbia, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
- San Jorge Children's Hospital, San Juan, Puerto Rico